CLINICAL TRIAL: NCT00825812
Title: A Multi-center, Randomized, Parallel-group, Active-controlled, Safety-assessor Blinded Trial, Comparing the Efficacy and Safety of 2.0 mg.Kg-1 Sugammadex With 50 μg.Kg-1 Neostigmine Administered at Reappearance of T2 After Rocuronium in Chinese and European ASA I-III Subjects Undergoing Elective Surgery Under Propofol Anesthesia
Brief Title: Comparison of 2.0 mg/kg Sugammadex and Neostigmine at Reappearance of T2 in Chinese and European Subjects (Study 19.4.324)(P05768AM1)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P05768; 19.4.324
Record Dates: First submitted 2009-01-15; First posted 2009-01-21 (Estimated); Results first posted 2011-08-18 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Anesthesia, General; Neuromuscular Blockade
MeSH Terms: interventions — Sugammadex; Neostigmine; Atropine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sugammadex in Caucasian Subjects (Experimental): At reappearance of T2 after the last dose of rocuronium, 2.0 mg.kg-1 sugammadex was administered.
  Interventions: Drug: Sugammadex
- Neostigmine in Caucasian Subjects (Active Comparator): At reappearance of T2 after the last dose of rocuronium, 50 μg.kg-1 neostigmine (combined with 10-20 μg.kg-1 atropine, in a ratio ranging from 2.5:1 to 5:1) was administered.
  Interventions: Drug: neostigmine
- Sugammadex in Chinese Subjects (Experimental): At reappearance of T2 after the last dose of rocuronium, 2.0 mg.kg-1 sugammadex was administered.
  Interventions: Drug: Sugammadex
- Neostigmine in Chinese Subjects (Active Comparator): At reappearance of T2 after the last dose of rocuronium, 50 μg.kg-1 neostigmine (combined with 10-20 μg.kg-1 atropine, in a ratio ranging from 2.5:1 to 5:1) was administered.
  Interventions: Drug: neostigmine

INTERVENTIONS:
Drug: Sugammadex — After induction of anesthesia an intubation dose of 0.6 mg/kg rocuronium was administered. Maintenance doses of 0.1-0.2 mg/kg rocuronium intravenous (IV) could be administered if necessary. At reappearance of T2 after the last administration of rocuronium, an IV single bolus dose of 2.0 mg/kg sugammadex was administered.
  Other Names: Org 25969, Bridion®
  Arms: Sugammadex in Caucasian Subjects; Sugammadex in Chinese Subjects
Drug: neostigmine — After induction of anesthesia an intubation dose of 0.6 mg/kg rocuronium was administered. Maintenance doses of 0.1-0.2 mg/kg rocuronium IV could be administered if necessary. At reappearance of T2 after the last administration of rocuronium, an IV single bolus dose of 50 µg/kg neostigmine (combined with 10-20 μg.kg-1 atropine, in a ratio ranging from 2.5:1 to 5:1) was administered.
  Other Names: Neostigmine with atropine
  Arms: Neostigmine in Caucasian Subjects; Neostigmine in Chinese Subjects

SUMMARY:
The present trial was set up to evaluate the efficacy and safety of 2.0 mg.kg-1 sugammadex compared to neostigmine administered at reappearance of T2 in Chinese and Caucasian subjects for registration purposes in China.

ELIGIBILITY:
Inclusion Criteria:

-Subjects who are willing to provide informed consent; be between 18 and 64 years old; are American Society of Anaesthesiology (ASA) class 1-3 (extremes included); scheduled for elective surgery under general anesthesia, allowing stable neuromuscular monitoring, which requires neuromuscular blockade using rocuronium; be compliant with the dose/visit schedules, and use an accepted method of contraception (if applicable).

For China only: Subjects of Chinese descent born in China, never emigrated out of China and have a Chinese home address. For Europe only: Subjects of Caucasian descent born in Europe, never emigrated out of Europe and have a European home address.

Exclusion Criteria:

-Subjects with expected difficult intubation, neuromuscular disorders affecting neuromuscular blockade, significant renal/hepatic dysfunction, use of a tourniquet, (family) history of malignant hyperthermia, allergy to general anesthesia medications, contraindication to study drugs, breast feeding, pregnant, participation in previous or new trials, a clinically significant condition that may interfere with the trial, or membership in the (family of) study/sponsor staff.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 308 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

REFERENCES:
- [Result] Wu X, Oerding H, Liu J, Vanacker B, Yao S, Dahl V, Xiong L, Claudius C, Yue Y, Huang Y, Abels E, Rietbergen H, Woo T. Rocuronium blockade reversal with sugammadex vs. neostigmine: randomized study in Chinese and Caucasian subjects. BMC Anesthesiol. 2014 Jul 12;14:53. doi: 10.1186/1471-2253-14-53. eCollection 2014. PMID 25187755

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 308 participants were randomized
Period: Overall Study
Arm/Group | Sugammadex in Caucasian Subjects | Neostigmine in Caucasian Subjects | Sugammadex in Chinese Subjects | Neostigmine in Chinese Subjects
Started | 29 | 32 | 126 | 121
TREATED | 29 | 31 | 120 | 111
Completed | 29 | 31 | 120 | 111
Not Completed | 0 | 1 | 6 | 10
Not completed — Never entered follow up | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Subject withdrew consent | 0 | 0 | 3 | 2
Not completed — Non-compliance with protocol | 0 | 0 | 0 | 1
Not completed — Administrative | 0 | 1 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex in Caucasian Subjects | Neostigmine in Caucasian Subjects | Sugammadex in Chinese Subjects | Neostigmine in Chinese Subjects | Total
Number analyzed (Participants) | 29 | 31 | 120 | 111 | 291
Age, Continuous [Mean (Full Range); unit: years] | 52.0 (10.3) [27 to 64] | 51.9 (7.3) [34 to 63] | 39.9 (10.8) [19 to 63] | 39.4 (10.8) [18 to 61] | 42.2 [18 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 28 | 78 | 86 | 217
  Male | 4 | 3 | 42 | 25 | 74

OUTCOME MEASURES:

1. Primary Outcome: Time From Start of Administration of Investigational Medicinal Product (IMP) to Recovery of the T4/T1 Ratio to 0.9.
Description: Neuromuscular functioning was monitored by applying repetitive train of four (TOF) electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. Nerve stimulation was to continue until the ratio of the magnitude of the fourth twitch (T4) to first twitch (T1) reached >= 0.9. The greater the T4/T1 ratio the greater the recovery from neuromuscular blockade, with a value of 1.0 representing full recovery.
  The primary analysis was the comparison between sugammadex & neostigmine among Chinese subjects; other comparisons were secondary.
Time Frame: start of administration of sugammadex/neostigmine to recovery from neuromuscular blockade
Population: The Full Analysis Set (FAS) population included all subjects who received randomized treatment and had at least one efficacy measurement. In the event of missing data, imputed data were used for analysis.
  291 subjects received IMP, of whom two had no efficacy measurements at all. Hence the FAS consisted of 289 subjects.
Measure: Geometric Mean (95% Confidence Interval); unit: minutes
Arm/Group | Sugammadex in Caucasian Subjects | Neostigmine in Caucasian Subjects | Sugammadex in Chinese Subjects | Neostigmine in Chinese Subjects
Number analyzed (Participants) | 29 | 30 | 119 | 111
minutes | 1.4 [1.3 to 1.5] | 6.7 [5.5 to 8.0] | 1.6 [1.5 to 1.7] | 9.1 [8.0 to 10.3]
Statistical Analysis 1: Comparison: Sugammadex in Chinese Subjects vs Neostigmine in Chinese Subjects; The primary analysis was the comparison of the two treatments among Chinese subjects; Test type: Superiority or Other; ANOVA; ANOVA, adjusted for center effects, on log transformed times from start of administration of IMP to recovery of the T4/T1 ratio to 0.9; ratio of geometric mean time to recovery = 5.7, 95% CI [4.9 to 6.6] — Ratio of time to recovery of 0.9 T4/T1 ratio (neostigmine time / sugammadex time)
Statistical Analysis 2: Comparison: Sugammadex in Caucasian Subjects vs Neostigmine in Caucasian Subjects; A key secondary analysis was the comparison of the two treatments among Caucasian subjects; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; ratio of geometric mean time to recovery = 4.8, 97.5% CI [3.7 to 6.0] — Ratio of time to recovery of 0.9 T4/T1 ratio (neostigmine time / sugammadex time)
Statistical Analysis 3: Comparison: Sugammadex in Caucasian Subjects vs Sugammadex in Chinese Subjects; A key secondary analysis was the comparison for equivalence between Chinese subjects and Caucasian subjects; Test type: Non-Inferiority or Equivalence — Equivalence was considered if the 97.5% confidence interval (CI) for median difference in recovery time (T4/T1 ratio to 0.9) was within the pre-specified range of -60 to +60 seconds; median difference (seconds) = 7, 97.5% CI [-5 to 21] — Estimated median difference (Chinese - Caucasian) in seconds for the time to recovery of the T4/T1 ratio to 0.9 (after sugammadex)

2. Secondary Outcome: Time From Start of Administration of IMP to Recovery of the T4/T1 Ratio to 0.7 and 0.8.
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. The greater the T4/T1 ratio the greater the recovery from neuromuscular blockade.
Time Frame: start of administration of sugammadex/neostigmine to recovery from neuromuscular blockade
Population: The Full Analysis Set population included all subjects who received randomized treatment and had at least one efficacy measurement. In the event of missing data, imputed data were used for analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: minutes
Arm/Group | Sugammadex in Caucasian Subjects | Neostigmine in Caucasian Subjects | Sugammadex in Chinese Subjects | Neostigmine in Chinese Subjects
Number analyzed (Participants) | 29 | 30 | 119 | 111
minutes
  Recovery of T4/T1 ratio to 0.7 | 1.0 [0.9 to 1.1] | 3.4 [3.0 to 3.8] | 1.1 [1.1 to 1.2] | 4.4 [4.0 to 4.9]
  Recovery of T4/T1 ratio to 0.8 | 1.2 [1.1 to 1.3] | 4.6 [4.0 to 5.4] | 1.3 [1.2 to 1.4] | 6.0 [5.4 to 6.7]

ADVERSE EVENTS:
Arm/Group | Sugammadex in Caucasian Subjects | Neostigmine in Caucasian Subjects | Sugammadex in Chinese Subjects | Neostigmine in Chinese Subjects
Serious Adverse Events (participants affected / at risk) | 0/29 | 2/31 | 0/120 | 1/111
Other Adverse Events (participants affected / at risk) | 18/29 | 26/31 | 73/120 | 84/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex in Caucasian Subjects (N=29) | Neostigmine in Caucasian Subjects (N=31) | Sugammadex in Chinese Subjects (N=120) | Neostigmine in Chinese Subjects (N=111)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex in Caucasian Subjects (N=29) | Neostigmine in Caucasian Subjects (N=31) | Sugammadex in Chinese Subjects (N=120) | Neostigmine in Chinese Subjects (N=111)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 6 (6) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 7 (9) | 10 (11) | 13 (13)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 11 (11) | 11 (11)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 16 (17) | 16 (16)
Sensation of foreign body (General disorders) | 0 (0) | 0 (0) | 8 (8) | 4 (4)
Anaesthetic complication cardiac (Injury, poisoning and procedural complications) | 0 (0) | 5 (5) | 1 (2) | 7 (7)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 28 (28) | 26 (26)
Procedural hypotension (Injury, poisoning and procedural complications) | 6 (8) | 14 (20) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 4 (4) | 7 (7)
Procedural pain (Injury, poisoning and procedural complications) | 13 (20) | 12 (15) | 10 (10) | 10 (10)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 4 (4) | 7 (7)
Wound complication (Injury, poisoning and procedural complications) | 3 (3) | 3 (4) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 11 (11) | 22 (23)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 5 (5) | 6 (6)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3) | 2 (2) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 5 (5) | 9 (9)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5) | 10 (10)
Hypotensive anaesthesia procedure (Surgical and medical procedures) | 1 (1) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI must not publish/publicly present any interim results without prior written consent of sponsor. The PI must provide copies of material for sponsor to review, 45 days prior to submission for publication/presentation. The sponsor may review/comment. If the parties disagree on the appropriateness of the data analysis and presentation, the PI must agree to meet prior to submission for publication/presentation to make good faith efforts to discuss and resolve any issues or disagreement.